CLINICAL TRIAL: NCT06430827
Title: Clinical Study of Irinotecan Hydrochloride Liposome Injection Combined With Capecitabine for Second-line Treatment in Patients With Advanced or Metastatic Biliary Tract Carcinoma.
Brief Title: Clinical Study of Irinotecan Hydrochloride Liposome Combined With Capecitabine for Second-line Treatment in Patients With Advanced or Metastatic Biliary Tract Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ba Yi (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Ba Yi, Director, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DNY-BTC-02
Record Dates: First submitted 2024-04-15; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Biliary Tract Carcinoma
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients will receive irinotecan hydrochloride liposome injection combined with Capecitabine therapy in a 2-week treatment cycle.
  Interventions: Drug: irinotecan hydrochloride liposome injection; Drug: Capecitabine

INTERVENTIONS:
Drug: irinotecan hydrochloride liposome injection — rinotecan hydrochloride liposome injection (70mg/m^2) will be administered by intravenous infusion on day 1 in a 2-week treatment cycle.
  Other Names: duoenyi
Drug: Capecitabine — Capecitabine (1000 mg/m^2) will be administered orally in a 2-week treatment cycle, twice a day from day 1 to day 10 of each cycle
  Other Names: Kapeitabin

SUMMARY:
To evaluate the efficacy and safety of irinotecan hydrochloride liposome injection combined with Capecitabine for second-line treatment in Patients With advanced or metastatic biliary tract carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient had good compliance, could understand the research process of this study, and signed a written informed consent.
2. Age ≥18 years.
3. Has histologically confirmed diagnosis of advanced (metastatic) and/or unresectable (locally advanced) biliary tract cancer (intra-or extrahepatic cholangiocarcinoma or gallbladder cancer).
4. Subjects who had received gemcitabine prior first-line therapy and had not received fluorouracil drugs.
5. Subjects who have progressed after receiving previous first-line therapy, relapse within 6 months after the end of (neo) adjuvant therapy is considered as first-line therapy failure.
6. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
7. ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.
8. Has a life expectancy of greater than 3 months.
9. LVEF≥50%.
10. Appropriate organ function is defined as follows: (Hematology and blood biochemistry tests must be completed within 14 days prior to enrollment, and the following criteria are met):

    1. ANC ≥1.5×10^9/L
    2. Hb≥90g/L
    3. PLT ≥100×10^9/L
    4. total bilirubin ≤1.5 x ULN
    5. ALT/AST ≤ 2.5 x ULN; When there is liver metastasis, ALT/AST ≤ 5 x ULN
    6. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr) ≥50mL/min (according to Cockcroft-Gault fórmula)
    7. Coagulation function: prothrombin time (PT), activated partial thromboplastin time (APTT) and international standardized ratio (INR) ≤1.5×ULN
11. Patients with biliary obstruction should receive adequate biliary drainage.
12. Adverse reactions caused by previous treatment must be restored to grade 1 or baseline according to CTCAE5.0 (except for toxicity such as alopecias, grade 2 and below peripheral neuropathy, which can be included after the investigator determines that there is no safety risk).
13. non-pregnant or lactating female; Effective contraception should be used by female/Male of childbearing age during the study period and for 6 months after the end of study treatment.
14. There were no contraindications for the use of irinotecan liposomes and capecitabine.

Exclusion Criteria:

1. Patients who have had other malignant tumors within the previous 5 years (except cured carcinoma in situ and skin basal cell carcinoma).
2. Uncontrolled pleural effusion or ascites.
3. Any known brain or meningeal metastases.
4. Subjects were co-administering a potent CYP3A4 inducer within 3 weeks prior to first dosing, or a potent CYP3A4 inhibitor or a potent UGT1A1 inhibitor within 3 weeks prior to first dosing.
5. Subjects underwent large organ surgery (except needle biopsy, central venous catheterization, port catheterization, stenting for relief of biliary obstruction, percutaneous hepatobiliary drainage, and cholecystostomy) or an elective surgical program within 4 weeks before the first dose of the study drug.
6. Active, uncontrolled bacterial, viral, or fungal infections with systemic treatment, defined as persistent signs/symptoms associated with infection that do not go away despite the use of appropriate antibiotics, antiviral therapy, and/or other treatment, including patients with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
7. Patients who are known to have dihydropyridine dehydrogenase (low activity) or deficiency.
8. There are serious concomitant diseases: such as uncontrolled diabetes after hypoglycemic drug treatment, uncontrolled hypertension, serious cardiovascular and cerebrovascular disease, kidney failure, liver failure, uncontrolled epilepsy, central nervous system disease or mental disorder history, clear gastrointestinal bleeding tendency, intestinal paralysis, intestinal obstruction, etc.
9. Grade 1 diarrhea with an increase in the number of stools > 4 times per day compared to baseline; The moderate and severe effluents from stoma increased; Limited activities of daily living with the aid of tools or even self-rational activities of daily living; Life-threatening; Need urgent medical attention.
10. Had participated in other clinical investigators within 4 weeks before enrollment.
11. Unsuitable for participation in the trial by the investigator assessed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | baseline up to approximately 6 months
  To evaluate the efficacy of anti-tumor

SECONDARY OUTCOMES:
Objective response rate (ORR) | baseline up to approximately 6 months
  To evaluate the efficacy of anti-tumor
Overall survival (OS) | baseline up to approximately 12 months
  To evaluate the efficacy of anti-tumor
Quality of life (QoL) | baseline up to approximately 12 months
  To identify the quality of life by QLQ-C30（V3.0）

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, Principal Investigator — PEKING UNION MEDICALCOLLEGE HOSPITAL
Locations (1):
- Peking Union Medicalcollege Hospital, Beijing, China